CLINICAL TRIAL: NCT04446598
Title: Non Ablative Erbium:YAG Laser Transurethral Treatment for Chronic Prostatitis/Chronic Pelvic Pain Syndrome in Younger Patients: a Prospective Comparative Study
Brief Title: Management of Prostatodynia in Younger Patients With Non-ablative Erbium:YAG Intraurethral Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adrian Gaspar (Other)
Responsible Party: Sponsor-Investigator, Adrian Gaspar, Principal Investigator, Espacio Gaspar Clinic
Organization: Espacio Gaspar Clinic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPPS/CP-01
Record Dates: First submitted 2020-06-03; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Chronic Prostatitis With Chronic Pelvic Pain Syndrome; Prostatodynia
MeSH Terms: conditions — Prostatitis | interventions — Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser group (Experimental): In the laser group, the patients received two sessions of Er:YAG intraurethral laser in non-ablative SMOOTH™ mode, with 1 month interval between sessions.
  Interventions: Device: non-ablative SMOOTH mode Erbium YAG laser
- Tadalafil group (Active Comparator): The tadalafil group was treated with daily oral administration of tadalafil, at a dose of 5 mg/day, which lasted consecutively for two months.
  Interventions: Drug: Tadalafil 5mg

INTERVENTIONS:
Device: non-ablative SMOOTH mode Erbium YAG laser — Erbium:YAG (Er:YAG) laser with non-ablative SMOOTH™ mode
  Arms: Laser group
Drug: Tadalafil 5mg — oral tadalafil 5 mg was administered daily over a period of two months
  Arms: Tadalafil group

SUMMARY:
This prospective study aimed to compare the clinical outcomes between the use of the erbium: YAG (Er:YAG) laser, intraurethrally administered in long non-ablative SMOOTH™ train of pulses applied at the level of the male prostatic urethra, to the use of the pharmacological treatment of oral tadalafil for the treatment of chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS). The results show that both treatments are effective in alleviating symptoms of CP/CPPS. The non-ablative Er:YAG SMOOTHTM laser seems to be a promising treatment for this widely spread condition. More studies are needed to confirm its safety and efficacy.

DETAILED DESCRIPTION:
Prostatitis is the most common diagnosis (>50%) in men visiting outpatient urological clinics .

The NIH classification classifies prostatitis into 4 types: category I - acute bacterial prostatitis, which is very rare, affecting only up to 5% of patients; category II- chronic bacterial prostatitis, also affecting up to 5% of patients; category III- chronic nonbacterial prostatitis/chronic pelvic pain syndrome (CP/CPPS), which is the most common, as it affects 90%-95% of cases; and Category IV- asymptomatic inﬂammatory prostatitis, which has unknown prevalence and also unknown clinical significance.

Although category III or CP/CPPS is the most prevalent form of prostatitis, its causes are largely unknown and treatments often fail to alleviate symptoms in the long term. In contrast, patients suffering from type I and II prostatitis are successfully treated with antibiotics, as a uropathogen or an infectious agent is usually identified as the cause .

CP/CPPS is characterized by pain in the perineum and tenderness in the prostate and various urological symptoms (urgency, frequency, low urethral pressure) and sometimes also ejaculatory symptoms, such as painful ejaculation.

Currently used treatments for CP/CPPS are mainly pharmacological, including alpha blockers, 5-alpha reductase inhibitors, anti-inflammatories, antibiotics, phytotherapy, allopurinol, botulinum toxin and traditional Chinese medicine . Non-pharmacological therapies include acupuncture, prostatic massage, extracorporeal shockwave therapy, pulsed magnetic field therapy, transrectal and transurethral thermotherapy and others . Some of the abovementioned therapies alleviate symptoms by improving vascularisation and blood flow of the prostate and peri-prostatic area. This is also the mechanism of action of the erbium:YAG (Er:YAG) laser with non-ablative SMOOTH™ mode - it works by thermal pulsing of the treated surface, with microsecond-range long pulses combined into long (several hundred millisecond range) sequences. Each laser micropulse sharply increases tissue temperature and acts as a stimulative trigger. Long pulse trains cause slower diffusion of heat to deeper layers of the skin or mucosa, causing initially vasodilation and then collagen remodelling and stimulation of fibroblasts with collagen remodelling. It has shown to improve vascularisation and alleviate symptoms of genitourinary syndrome of menopause (GSM) in women, including irritation, dryness and pain. It has also been used intraurethrally in women to alleviate urinary symptoms of GSM. Intraurethral thermal therapy has been previously shown promising in the treatment of CP/CPPS in men. In this study the investigators aimed to assess the safety and effectiveness of transurethral non-ablative Er:YAG laser therapy applied at the level of the male prostatic urethra and to compare it with pharmacological treatment of 5 mg oral tadalafil for the treatment of CP/CPPS.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of chronic prostatitis/chronic pelvic pain syndrome with characteristic symptoms of perineal pain and urinary symptoms of dysuria and urinary frequency;
* negative urine culture after prostatic massage; prostatic volume less than 50 cc in prostatic ultrasound;
* obstructive uroflowmetric pattern with a Q-max value between 10 and 15 ml/sec

Exclusion Criteria:

* age over 50 years
* current or recent (last 6 months) pharmacological or other therapies of CP/CPPS

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum urethral flow value (Q-max) | Change from Baseline Q-max at 3 and 6 months following the intervention
  measurement of maximum urethral flow using uroflowmetry
IPSS questionnaire | Change from Baseline IPSS score at 1, 3, 6 and 12 months following the intervention
  Assessment of urinary symptoms using the International Prostate Symptom Score (IPSS)

SECONDARY OUTCOMES:
pain assesment: VAS (visual analog scale) scale | Change from Baseline pain VAS score at 1, 3, 6 and 12 months following the intervention
  subjective assesment of pain using 0 (minimum) to 10 (maximum) VAS scale. 0 means no pain, 10 means worst possible pain;
dysuria assesment: VAS (visual analog scale) scale | Change from Baseline dysuria VAS score at 1,3, 6 and 12 months following the intervention
  subjective assesment of dysuria using 0 (minimum) to 10 (maximum) VAS scale. 0 means no dysuria, 10 means worst possible dysuria;
Patient satisfaction: 7-point Likert Scale | 6 months following the intervention
  subjective assessment of patients' satisfaction with the treatment using 0 to 6 Likert Scale; Question - How satisfied are you with the treatment? Likert scale: 0 - extremely satisfied; 1- very satisfied; 2 - mostly satisfied; 3 - neither satisfied nor unsatisfied; 4 - mostly unsatisfied; 5 - very unsatisfied; 6- extremely unsatisfied
Patient satisfaction: 7-point Likert Scale | 12 months following the intervention
  subjective assessment of patients' satisfaction with the treatment using 0 to 6 Likert Scale; Question - How satisfied are you with the treatment? Likert scale: 0 - extremely satisfied; 1- very satisfied; 2 - mostly satisfied; 3 - neither satisfied nor unsatisfied; 4 - mostly unsatisfied; 5 - very unsatisfied; 6- extremely unsatisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Uroclinica, Mendoza, Argentina

IPD SHARING:
Plan to Share IPD: No